CLINICAL TRIAL: NCT04612023
Title: A Prospective, Double-Blinded, Randomized Controlled Trial of an Amniotic Membrane Allograft Injection Comparing Two Doses (1 mL and 2mL Injection) and a Placebo (Sterile Saline) in the Treatment of Osteoarthritis of the Knee
Brief Title: An Amniotic Membrane Injection Comparing Two Doses (1 mL and 2 mL Injection) and a Placebo (Sterile Saline) in the Treatment of Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Illinois Center for Orthopaedic Research and Education (Other)
Responsible Party: Principal Investigator, Eyal Ginesin, Orthopedic Surgeon / Fellow Researcher, Illinois Center for Orthopaedic Research and Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8212
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; amniotic fluid; amniotic allograft; knee; amniotic membrane
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Data will be prospectively collected on all injectable acellular amniotic membrane derived allograft knee performed at our institute. (FDA regulated - HCT/P regulation)
  Inclusion criteria will be all patients age between 21 and 80 years with a diagnosis of osteoarthritis (OA) defined as Grade 1 to 3 on the Kellgren Lawrence grading scale.
  Methods for collecting data will be through validated patient-reported outcome tools that the patient will complete pre-injection and at specified time intervals after injection: 30 days, 90 days, 180 days and 365 days.
  Patient will receive a phone call 24 hours after the injection to monitor any immediate potential adverse events.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Assistants not part of the study used a randomizer generating software to randomly assign a patient a dose. The randomly assigned dose was put in a sealed envelope labeled with the corresponding number and was recorded. Prior to the injection, a medical assistant not involved in the study retrieves the envelope to determine the dose, prepares the injection, then seals the syringe in black tape before giving it to the research staff who then performs the injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 mL NyDYN Injection (Active Comparator): 30 patients (out of 90) will be blind to and randomly assigned to a 1 mL NyDYN injection.
  Interventions: Other: Acellular Amniotic Membrane Derived Allograft Injection (NuDYN)
- 2 mL NuDYN Injection (Active Comparator): 30 patients (out of 90) will be blind to and randomly assigned to a 2 mL NyDYN injection.
  Interventions: Other: Acellular Amniotic Membrane Derived Allograft Injection (NuDYN)
- Placebo of Sterile Saline (Placebo Comparator): 30 patients (out of 90) will be blind to and randomly assigned to a 2 mL dose of sterile saline.
  Interventions: Other: Acellular Amniotic Membrane Derived Allograft Injection (NuDYN)

INTERVENTIONS:
Other: Acellular Amniotic Membrane Derived Allograft Injection (NuDYN) — Injectable acellular amniotic membrane derived allograft tissue (NuDYN) through routine follow-up with physical examination, pain, function and quality of life measurements and compare dose effects (1 mL versus 2 mL of NuDYN injection) to a placebo (sterile saline) in the treatment of knee osteoarthritis. Injection is minimally invasive and is FDA regulated (HCT/P regulation).

SUMMARY:
The purpose of this study is to determine the dose effect of a single injectable acellular amniotic membrane derived allograft for the treatment of knee osteoarthritis and to confirm whether the use of 2 mL of the same amniotic injection offers a statistically significant advantage over the 1 mL injection when compared to a placebo.

DETAILED DESCRIPTION:
It is a prospective, double blinded, Randomized Controlled Trial study. Data will be prospectively collected of all injectable acellular amniotic membrane derived allograft knee performed at our institute (1 vs 2 mL).

90 subjects will be enrolled in the study. Subjects will be randomized 1:1:1 in treatment arms.

It compares the dose affect of an amniotic membrane allograft between a 1 mL dose and a 2 mL dose when compared to a placebo of sterile saline in the treatment of osteoarthritis of the knee. This will be offered as a free pain management alternative to patients who meet the inclusion criteria. The results will be determined by validated patient-reported outcome tools (KOOS, VAS, and WOMAC questionnaires) and physical examinations taken before the injection, one month after the injection, three months after the injection, six months after the injection, and one year after the injection. There will be a phone call 24 hours after the injection for every patient participating in the study regarding any potential adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for non-surgical intervention of the knee
* Patient must be between the ages of 21 and 80 years old
* Patient must have a diagnosis of osteoarthritis (OA) of the knee defined as grade 1 to 3 on the Kellgren-Lawrence grading scale

Exclusion Criteria:

* Patient has a diagnosis of osteoarthritis with a Kellgren-Lawrence grade of 4
* Patient has a BMI greater than 40 kg/m2, active infection at the injection site, symptomatic OA of the contralateral knee or of either hip that is not responsive to acetaminophen (Tylenol) and requires other therapy
* Patient has rheumatoid arthritis, psoriatic arthritis or diagnosis with any other disorder that is the primary source of their knee pain
* Patient has an autoimmune disease or known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV
* Patient has any of the following treatments to the target knee within 12 weeks prior to screening
* Intra-articular hyaluronic acid (HA) injection
* Steroid or platelet rich plasma (PRP) injection
* Use of any investigational drug, device, or biologic
* Patient had or is planning to have major surgery or arthroscopy in the target knee within 26 weeks of treatment
* Patient has a history of partial or total knee arthroplasty
* Patient has undergone immunotherapy or chemotherapy in the last 5 years, prior radiation at the site, or is currently taking a narcotic medication for any reason
* Patient is pregnant or plans to become pregnant within 365 days of treatment
* Patient has any significant medical condition that would interfere with protocol evaluation and participation
* Patient is a recipient of worker's compensation
* Patient is a current prisoner

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-04-02 (Estimated); Study Completion 2022-07-02 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoints using Validated patient-reported outcome tools questionnaires | 1 year
  Knee injury and Osteoarthritis Outcome Score (KOOS)- assess five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. It is a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Primary Efficacy Endpoints using Validated patient-reported outcome tools questionnaires | 1 year
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)- assess the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. it is a 0 (worst)-96 scale (best).
Primary Efficacy Endpoints using Validated patient-reported outcome tools questionnaires | 1 year
  Visual Analogue Scale (VAS)- assess pain, It is a 0-100 scale. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Exploratory Endpoint using Validated patient-reported outcome tools questionnaires | 30, 90, 180, 365 days
  Change from baseline Knee injury and Osteoarthritis Outcome Score (KOOS)- assess five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. It is a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Exploratory Endpoint using Validated patient-reported outcome tools questionnaires | 30, 90, 180, 365 days
  Change from baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)- assess the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. it is a 0 (worst)-96 scale (best).
Exploratory Endpoint using Validated patient-reported outcome tools questionnaires | 30, 90, 180, 365 days
  Change from baseline Visual Analogue Scale (VAS)- assess pain, It is a 0-100 scale. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Nikil Chari, Study Chair — Research Assistant; Jacob Barnhart, Study Chair — Research Assistant
Locations (1):
- ICORE, Westmont, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riboh JC, Saltzman BM, Yanke AB, Cole BJ. Human Amniotic Membrane-Derived Products in Sports Medicine: Basic Science, Early Results, and Potential Clinical Applications. Am J Sports Med. 2016 Sep;44(9):2425-34. doi: 10.1177/0363546515612750. Epub 2015 Nov 19. PMID 26585668
- [Background] Vines JB, Aliprantis AO, Gomoll AH, Farr J. Cryopreserved Amniotic Suspension for the Treatment of Knee Osteoarthritis. J Knee Surg. 2016 Aug;29(6):443-50. doi: 10.1055/s-0035-1569481. Epub 2015 Dec 18. PMID 26683979